CLINICAL TRIAL: NCT02359331
Title: A Prospective, Single-center, Randomized, Open-label, Parallel Design Clinical Trial to Compare the 14-day Bismuth Quadruple Therapy and 7-day Culture Based Tailored Therapy for the Eradication of Helicobacter as a Rescue 2nd Therapy.
Brief Title: The Efficacy of the 7 Days Tailored Therapy as 2nd Rescue Therapy for Eradication of H. Pylori Infection
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Nayoung Kim, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B1408/285-005
Record Dates: First submitted 2015-02-04; First posted 2015-02-10 (Estimated); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Helicobacter Infection
Keywords: Helicobacter pylori; resistance; rescue therapy
MeSH Terms: conditions — Helicobacter Infections | interventions — Proton Pump Inhibitors; Metronidazole; Tetracycline; Moxifloxacin; Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 14 days PBMT group (Active Comparator): Giving the 14 days bismuth quadruple regimen as 2nd rescue therapy for eradication of persistent H. pylori infection Drug regimen Proton pump inhibitor (PPI) regular dose b.i.d., tripotassium dicitrate bismuthate 300 mg q.i.d. (three tablets at 30 min before meals and one tablet at 2 hours after dinner), metronidazole 500 mg t.i.d., and tetracycline 500 mg q.i.d
  Interventions: Drug: 14 days empirical bismuth quadruple therapy (Proton pump inhibitor); Drug: Metronidazole; Drug: Tetracycline; Drug: tripotassium dicitrate bismuthate
- 7 days tailored therapy group (Experimental): According the antimicrobial susceptibility testing, the H. pylori isolates were resistant to moxifloxacin, 7 days PBMT regimen were prescribed; if the isolates were resistant to metronidazole, 7 days moxiflxacin based triple regimen (PPI regular dose b.i.d., moxifloxacin 400 mg q.d., and amoxicillin 1g b.i.d) were prescribed.
  Interventions: Procedure: H. pylori culture and antimicrobial susceptibility testing; Drug: 7 days tailored therapy Proton Pump Inhibitor; Drug: Moxifloxacin; Drug: Amoxicillin

INTERVENTIONS:
Procedure: H. pylori culture and antimicrobial susceptibility testing — This intervention will be performed in 7 days tailored therapy group.
  All the patients who enrolled in this arm, they will be received endoscopy guided biopsy procedure. Minimum inhibitory concentrations (MICs) were determined by the agar dilution method. Amoxicillin, clarithromycin, metronidazo, tetracycline and moxifloxacin for the H. pylori isolates were examined by use of the serial two fold agar dilution method
  Arms: 7 days tailored therapy group
Drug: 14 days empirical bismuth quadruple therapy (Proton pump inhibitor) — Giving the 14 days PBMT regimen as 2nd rescue therapy
  Proton pump inhibitor (PPI) regular dose b.i.d., tripotassium dicitrate bismuthate 300 mg q.i.d. (three tablets at 30 min before meals and one tablet at 2 hours after dinner), metronidazole 500 mg t.i.d., and tetracycline 500 mg q.i.d.
  Arms: 14 days PBMT group
Drug: Metronidazole
  Arms: 14 days PBMT group
Drug: Tetracycline
  Arms: 14 days PBMT group
Drug: tripotassium dicitrate bismuthate
  Arms: 14 days PBMT group
Drug: 7 days tailored therapy Proton Pump Inhibitor
  Arms: 7 days tailored therapy group
Drug: Moxifloxacin
  Arms: 7 days tailored therapy group
Drug: Amoxicillin
  Arms: 7 days tailored therapy group

SUMMARY:
As increasing the antibiotics resistance, the effectiveness of traditional Helicobacter pylori (H. pylori) therapies has been declined coincidentally.

In this study, the investigators evaluated the efficacy of H. pylori eradication between a 7 days personalized therapy for H. pylori infection based on the results of antibiotics resistance by using H. pylori culture and minimal inhibitory concentration (MIC) and the 14 days bismuth contained quadruple 2nd rescue regimens, and the investigators analyzed the prevalence of the antibiotic resistance after 1st eradication of H. pylori in the tailored therapy group.

DETAILED DESCRIPTION:
The patients who had shown the evidence of persistent H. pylori infection after the 1st eradication were enrolled for this study.

After giving the informed consent about the method and efficacy (ITT and PP analysis) of the 14 days bismuth quadruple 2nd rescue therapy and the 7 days tailored therapy for H. pylori infection based on culture and MIC, the patients were randomly classified into the two regimen group under the patient's agreement and underwent 2nd eradication [14 days bismuth-based quadruple therapy (Proton pump inhibitor (PPI) regular dose b.i.d., tripotassium dicitrate bismuthate 300 mg q.i.d. (three tablets at 30 min before meals and one tablet at 2 hours after dinner), metronidazole 500 mg t.i.d., and tetracycline 500 mg q.i.d.), or 7 days tailored therapy based on H. pylori culture and MIC (select the 2nd rescue regimen between 7 days of bismuth-based quadruple therapy or 7 days moxifloxacin-containing triple therapy (PPI regular dose b.i.d., moxifloxacin 400 mg q.d., and amoxicillin 1g b.i.d.) according to antibiotics susceptibility.

This study was designed to evaluate the success of eradication for enrolled participants by methods of an open labelled randomized prospectively.

ELIGIBILITY:
Inclusion Criteria:

* The patients who proved a failure of 1st eradication of H. pylori with Proton pump inhibitor based triple therapy (PPI bid + amoxacillin 1g b.i.d + Clarithromycin 500 mg b.i.d) or sequential therapy (initial 5-day therapy with a combination of PPI b.i.d and amoxicillin 1g b.i.d, followed by 5 days of PPI b.i.d., clarithromycin 500mg b.i.d., and metronidazole 500mg t.i.d) following three methods

  1. positive rapid urease test (CLOtest)
  2. histologic evidence of H. pylori by modified Giemsa staining
  3. positive 13C-Urea breath test
* Male and female Korean Adult (Aged ≥ 18 years)

Exclusion Criteria:

* Patients who received two or more eradication therapy for H. pylori infection
* H. pylori eradication failure because of poor compliance
* the administration of antibiotics or the consumption of bismuth salts within 4 weeks or the administration of a proton pump inhibitor (PPI) within 2 weeks
* Advanced gastric cancer or other malignancy
* Abnormal liver function or liver cirrhosis
* Abnormal renal function or chronic kidney disease
* Other severe concurrent diseases
* Previous allergic reactions to the study drugs
* Pregnant or lactating women

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2014-08; Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Compare the percentage of participants with successful H. pylori eradication in each groups | 6 weeks after completion of eradication
  The efficacy of H. pylori eradication between a 7 days tailored therapy for H. pylori infection based on the results of antimicrobial resistance by using H. pylori culture and minimal inhibitory concentration (MIC) and the 14 days bismuth quadruple therapy as 2nd rescue regimens.
  The eradication rate was evaluated by intention to treat (ITT) and per-protocol (PP) analysis

CONTACTS AND LOCATIONS:
Overall Officials: Nayoung Kim, M.D., Ph. D, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea